CLINICAL TRIAL: NCT03503825
Title: A Phase 1, Open-label, Non-Randomized Study to Evaluate the Safety and Tolerability of [Tc-99m]-RPI T-087 Injection as an Imaging Marker for COX-2 in Subjects With Osteoarthritis of the Knee Compared to Healthy Volunteers
Brief Title: [Tc-99m]-RPI-087 as an Imaging Marker in Osteoarthritis of the Knee Compared to Healthy Volunteers
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Reiley Pharmaceuticals Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: RPI-T-087-001
Record Dates: First submitted 2018-04-06; First posted 2018-04-20 (Actual); Last update posted 2019-01-15 (Actual); Status verified 2019-01

CONDITIONS: Healthy; Osteo Arthritis Knee

STUDY DESIGN:
Intervention Model Description: This is a Phase 1, non-randomized, open-label, single-centre clinical trial. A total of 12 to 24 subjects will be enrolled:
  * 6 Healthy volunteers (HV) (3 males and 3 females)
  * 6 - 18 subjects with osteoarthritis of the knee (KOA) Once 6 HVs and 6 KOA subjects (to be enrolled concurrently) have completed the study, image data will be assessed to determine whether any more KOA subjects should be imaged.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Healthy Volunteers (Experimental): Healthy volunteers will be administered [Tc-99m]-RPI-T-087 Injection, single IV dose of 555 MBq and will be monitored for safety, knee image evaluation, and radioactivity biodistribution and dosimetry.
  Interventions: Drug: [Tc-99m]-RPI-T-087 Injection
- Osteo Arthritis of the knee (Experimental): Subjects with knee osteoarthritis will be administered [Tc-99m]-RPI-T-087 Injection, single IV dose of 555 MBq and will be monitored for safety and knee image evaluation.
  Interventions: Drug: [Tc-99m]-RPI-T-087 Injection

INTERVENTIONS:
Drug: [Tc-99m]-RPI-T-087 Injection — A single intravenous injection of [Tc-99m]-RPI-T-087 followed by SPECT/CT imaging of the knee (all subjects) and whole body planar imaging (Healthy volunteers only)
  Other Names: T-087

SUMMARY:
The main purpose of this study is to test the safety and tolerability of T-087. The study will enroll 6 healthy volunteers (HVs) and 6-18 subjects with KOA. All eligible subjects will receive an intravenous injection of the radioactive investigational product (ip) (T-087), followed by SPECT/CT imaging of the knees and blood tests and clinical assessments for safety monitoring. Healthy volunteers will also have their whole body imaged and have extra blood drawn to determine where T-087 goes in the body. These additional procedures will be done on the same day as the ip administration, and repeated the following day. All subjects will have a final follow-up phone call within 2- 3 business days following the ip administration.

DETAILED DESCRIPTION:
This is a Phase 1, non-randomized, open label, single centre clinical trial. 6 healthy volunteers (3 male and 3 female,4 study visits) and 6-18 subjects with Osteoarthritis of the knee (3 study visits) will be enrolled. At visit 2, all subjects will have knee pain assessed, using a visual analogue scale, prior to receiving a single, 555 MBq (15 mCi)+/-10% dose of [Tc-99m)-RPI-T-087 injection. Knees will be imaged with a SPECT/CT camera at specified time-points post injection. Safety monitoring will include vital signs, ECG, clinical laboratory tests (serum biochemistry, haematology, urinalysis) and adverse event monitoring.

Additionally, HVs will have whole body planar imaging and blood sampling conducted at Visit 2 and 3 to evaluate bio-distribution, estimate dosimetry and measure clearance of total activity over time in blood samples. A final follow-up visit will be conducted by phone interview.

Once 6 HVs and 6 KOA participants have completed the study, a blinded assessment of the image data will be conducted to determine whether any more KOA subjects should be imaged.

ELIGIBILITY:
Inclusion Criteria :

* All subjects must be able to read and speak in English and capable of giving signed informed consent.
* Female subjects must either, not be of reproductive potential, or not be pregnant and be willing to comply with appropriate family planning methods as specified in the protocol.
* Male subjects must either, not be of reproductive potential or be willing to comply with appropriate family planning methods as specified in the protocol.

Subjects with Knee Osteoarthritis (KOA)

* Age ≥ 40 to ≤ 70 years, at the time of signing the informed consent
* Have chronic pain due to OA of at least one knee identifiable as the target knee as their primary pain condition and some degree of pain every day from this condition.

For Healthy Volunteers:

* Age ≥ 18 to ≤ 35 years, at the time of signing the informed consent.
* No history of knee pain or known knee pathology confirmed by knee radiographs, obtained within the last year.

Exclusion Criteria:

* Chronic pain conditions other than OA of the knee (KOA) as their predominant pain condition
* Cannot or will not agree to stop: all topical, oral and parenteral non-steroidal anti-inflammatory drugs (NSAIDs) for at least 48 hours before administration of the IP; stop turmeric and curcumin (supplements and dietary sources) for at least 48 hours before administration of the IP; avoid all exercise from at least 24 hours before administration of the IP up to the end of the last applicable imaging session.
* Systemic (including inhaled) and oral corticosteroid use currently or within 6 weeks prior to Visit 1.
* Surgical interventions of either knee or any other major surgery within the previous 6 months.
* Receipt of intra-articular corticosteroid injections within the previous 6 weeks prior to Visit 1 in the target knee or within the previous 2 weeks prior to Visit 1 in any other joint.
* Use of any other investigational medication or devices within 30 days prior to Visit 1.
* Orthopedic or prosthetic appliance in either knee which may confound scan interpretation.
* Screening ECG or laboratory assessments showing clinically significant abnormalities
* Refusal or inability to tolerate the scanning procedures
* Allergies to or cannot tolerate NSAIDs, the investigational product or sulfa drugs
* History of bleeding disorders or history of documented gastrointestinal ulcer disease.
* Received significant ionizing radiation exposure, in the last 12 months or undergoing occupational monitoring for radiation exposure.
* Allergies or sensitivity to any component of the investigational product. Subjects taking disulfiram (Antabuse) should be excluded from this study.
* History of alcohol or substance abuse
* Any medical condition or disease that in the opinion of the investigator makes the subject unsuitable to participate in this study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2018-08-16 (Actual); Primary Completion 2019-05-31 (Estimated); Study Completion 2019-06-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of treatment emergent adverse events | Up to 3 days post investigative product administration
  The incidence of adverse events, including injection site reactions, clinically significant changes in clinical laboratory parameters (blood and urine), ECG's and vital signs, will be summarized over time to assess safety and tolerability.

SECONDARY OUTCOMES:
Uptake over time | Up to 4.5 hours post administration of the investigational product
  Quantitative standard uptake values (SUV) for T-087 will be determined for the knees of subjects with KOA and HVs, and comparing uptake in the target knee of OA subjects with the uptake in the knees of the HVs.
Image quality | Up to 4.5 hours post administration of the investigational product
  A visual assessment using a scoring system will be used to assess the SPECT/CT images quality in subjects with KOA. Image quality scales of 1 to 3, with 1 as unacceptable (non-interpretable quality), 2 as adequate quality for interpretation and 3 as excellent quality (no issues) of the target knee will be descriptively summarized by time point and subject group.
Dosimetry | Up to 1 day post administration of the investigational product.
  Whole body planar imaging of healthy volunteers will be used to evaluate the biodistribution of [Tc-99m]-RPI-T-087 Injection to estimate dosimetry. Whole body scintigraphic images will be quantified as to fractional activity (IA) in various visceral organs (e.g., liver, lungs, heart) as well as routes of excretion, total body and knees. The data describing the uptake, retention and clearance in these tissues will characterize the biodistribution and biokinetics of the IP. These data also serve as the foundation for radiation dose estimates for the IP.

OTHER OUTCOMES:
Clearance of [Tc-99m]-RPI-T-087 | Up to 1 day post administration of the investigational product.
  Blood sampling (HVs only) will support the exploratory objective of using radioactivity measurements (if measurable) to assess the clearance of [Tc-99m]-RPI-T-087.

CONTACTS AND LOCATIONS:
Overall Officials: Karen Gulenchyn, MD, Principal Investigator — St. Joseph's Hospital Hamilton
Locations (1):
- St. Joseph's Healthcare Hamilton, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No